CLINICAL TRIAL: NCT05618860
Title: Patient Perspectives on Artificial Intelligence in Radiology
Acronym: PPAIR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 312778
Record Dates: First submitted 2022-10-27; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Patients Waiting for Radiology Exams
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — eligible participants in the radiology department waiting rooms will be asked to complete a questionnaire after taking consent.

SUMMARY:
The investigators will conduct a short questionnaire with patients who are waiting for radiology exams to understand their views on the use of artificial intelligence in radiology. The questionnaire will be anonymised and entirely optional. Results will be published in peer-reviewed publications and inform future implementation of AI in clinical radiology.

DETAILED DESCRIPTION:
The project entails a patient questionnaire. Patients will firstly be informed about the study via a member of the radiology care team. Informed consent will be obtained by a member of the team. Each participant will be assigned a unique identifier number upon recruitment. Aside from the signed consent form, no identifiable information or medical details will be collected. Consent documentation will be stored within a locked drawer in the research department of the radiology department in GSTT. The signed consent document will be kept entirely separate and will not be linked in any way to the questionnaire answers. The questionnaire data will therefore be anonymised data. A document containing the following items will be created on a GSTT computer and updated as the study progresses:

1. Participant Unique Identifier
2. Questionnaire Answers 5.2 Questionnaire When the study identifier number is assigned, it will be entered at the top of a paper questionnaire. The questionnaire is thus anonymised from the beginning of the study. The questionnaire will include demographic variables and questions with multiple choice responses corresponding to a Likert scale, which will be completed by the patient. This information will be transferred to an NHS computer in the radiology department in GSTT.

Survey data will not include identifiable information. A Gaussian Graphical Model will be inferred indicating conditional dependencies between demographic variables and participant responses. This will be performed using the desparsified Graphical LASSO method of Jankova, implemented via the R package SILGGM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to the radiology department waiting area for an elective appointment will be eligible to participate.
2. Participants must be aged above 18 years.
3. Participants must have independent capacity to consent to the study.

Exclusion Criteria:

1. Inpatients or acute patients presenting to the radiology department waiting area.
2. Those who cannot complete informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the radiology department waiting area for an elective appointment
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
This study aims to evaluate patient opinion regarding the use of artificial intelligence in radiology by completing a questionnaire | 6 months
  We aim to identify common concerns held by patients and to characterise the distribution of patient viewpoints regarding the use of artificial intelligence for radiology.This will allow identification of key issues from the patients' perspectives

SECONDARY OUTCOMES:
Quantification of patients' positivity towards AI technology in radiology by completing a questionnaire | 6 months
  This will facilitate understanding between expert and lay stakeholders on this issue.

IPD SHARING:
Plan to Share IPD: Undecided